CLINICAL TRIAL: NCT01674777
Title: A Pharmacokinetic Study to Investigate the Effect of Food on the Pharmacokinetics of ASP1941
Brief Title: A Study to Investigate the Effect of Food on the Absorption, Distribution and Elimination of ASP1941
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1941-CL-0071
Record Dates: First submitted 2012-08-21; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Healthy; Pharmacokinetics of ASP1941
Keywords: ASP1941; Food effect; Pharmacokinetics
MeSH Terms: interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- under fasting condition group (Experimental): Subjects will receive a single dose of ASP1941 under fasting condition
  Interventions: Drug: ASP1941
- before meal group (Experimental): Subjects will receive a single dose of ASP1941 before meal
  Interventions: Drug: ASP1941
- after meal condition (Experimental): Subjects will receive a single dose of ASP1941 after meal
  Interventions: Drug: ASP1941

INTERVENTIONS:
Drug: ASP1941 — oral
  Other Names: ipragliflozin

SUMMARY:
This study is to investigate the effect of food on the pharmacokinetics, the pharmacodynamics and safety of ASP1941 after administration of ASP1941 in healthy non-elderly adult male subjects.

DETAILED DESCRIPTION:
This will be a randomized, open-label, 3-way crossover design study to investigate the effect of food on the pharmacokinetics, the pharmacodynamics and safety of ASP1941 after administration of ASP1941 in healthy non-elderly adult male subjects. Each subject will receive a single dose of ASP1941 "under fasting condition", "before meal" and "after meal".

ELIGIBILITY:
Inclusion Criteria:

* Healthy as judged by the investigator/subinvestigator based on the results of physical examinations and laboratory tests
* Body weight ; ≥50.0 kg, <80.0 kg
* Body Mass Index ; ≥17.6, <26.4
* Written informed consent has been obtained

Exclusion Criteria:

* Received any investigational drugs within 120 days before the screening assessment
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or d components within 14 days before the screening assessment
* Received medication within 7 days before hospital admission
* A deviation from the assessment criteria of physical examinations or laboratory tests at screening or upon admission
* History of drug allergies
* With renal, hepatic, gastrointestinal, heart, cerebrovascular or respiratory diseases

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) profiles of ASP1941 (in plasma): AUCinf, AUClast and Cmax | For 72 hours after each administration
  Area under the curve (AUC) from time 0 extrapolated to infinity (AUCinf), AUC from time of dosing to last quantifiable concentration (AUClast ), and maximum concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) profiles of ASP1941 (in plasma): tmax, t1/2, apparent distribution volume, apparent body clearance | For 72 hours after each administration
  Time to attain Cmax (tmax) , apparent terminal elimination half-life (t1/2 )
Safety assessed by incidence of adverse event, vital signs, 12-lead ECG and laboratory tests | For 72 hours after each administration
Changes in urinary glucose excretion | Before and for 72 hours after each administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan